CLINICAL TRIAL: NCT01094574
Title: Investigation of Analgesic and Anti-inflammatory Effects of Beta-adrenergic Antagonist Propranolol
Brief Title: Evaluation of Propranolol's Effect on Pain and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Angst (Other)
Responsible Party: Sponsor-Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SU-10012009-4121; 17743
Record Dates: First submitted 2010-03-02; First posted 2010-03-29 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Pain Measurement
MeSH Terms: interventions — Alfentanil; Propranolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alfentanil (Active Comparator): Experimental inflammation, and tissue injury sites were created, an infusion of alfentanil 100ng/ml was administered over 3 hours using a programmable infusion pump, and data were collected to measure inflammation, pain response, and cytokine levels locally.
  Interventions: Drug: Alfentanil
- Propranolol (Active Comparator): Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours using a programmable infusion pump, and data were collected to measure inflammation, pain response, and cytokine levels locally.
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump, and data were collected to measure inflammation, pain response, and cytokine levels locally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alfentanil — An infusion of alfentanil 100ng/ml was administered over 3 hours using a programmable infusion pump.
  Other Names: No other name
  Arms: Alfentanil
Drug: Propranolol — An infusion of propranolol 30ng/ml was administered over 3 hours using a programmable infusion pump.
  Other Names: No other name
  Arms: Propranolol
Drug: Placebo — An infusion of normal saline was administered over 3 hours using a programmable infusion pump to mimic the 2 drug arms,
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Previous studies have shown that the beta-adrenergic system plays a role in processing pain and the expression of hyperalgesia. Recent studies have investigated the analgesic effects, and potential anti-hyperalgesic effects (using a model of opioid induced (OIH) hyperalgesia) of propranolol, a beta adrenergic antagonist. We plan to further investigate the analgesic effects, and the potential anti inflammatory effects, of propranolol and compare those effects to alfentanil, an opioid of known effect, and placebo

DETAILED DESCRIPTION:
This study is a double blind-placebo controlled study in which subjects will be exposed to propranolol infusion during one study day, the opioid alfentanil on another day, and placebo infusion during a third study day. The infusion order will be randomized, and the participant and individual conducting the pain testing will both be blinded to the treatment.

Propranolol, alfentanil, and placebo infusions will be administered intravenously using a computer-controlled infusion pump that can be set to accurately administer a target plasma concentration of drug.

On one study day subjects will receive propranolol at a target concentration of 30ng/ml over 3 hours time. On another study day subjects will receive 100ng/ml alfentanil over 3 hours, and on a third study day subjects will receive placebo (normal saline) using a computer-controlled infusion paradigm.

Sites to be evaluated for response to propranolol and placebo will be established in 2 ways. One will use ultraviolet B (UVB) exposure to create a "sunburn" causing inflammation and pain. The other will be a model of acute injury using an array of micro-needles.

Means of evaluation of injured, and non-injured sites will be pain testing (heat and mechanical pain thresholds will be established), interstitial fluid sampling for detection of pro-inflammatory, and pro-nociceptive cytokines, and laser doppler evaluation of tissue perfusion.

Subjects will be recruited using flyers. Interested participants will contact the study team, their questions will be answered, and an appointment for screening will be made.

ELIGIBILITY:
Inclusion Criteria:1) Age 18-65 2) Skin type II-IV according to classification of Fitzpatrick 3) Willing and able to sign an informed consent form and Health Insurance Portability and Accountability Act (HIPAA) authorization and to comply with study procedures

Exclusion Criteria:1) History of acute or chronic illness that contraindicate the use of propranolol, may hinder study procedures, or confuse interpretation of the data (e.g. cardiac, dermatological, neurological, psychiatric or addictive diseases) 2) Clinically significant cardiovascular, pulmonary, hepatic or renal diseases 3) Pregnant or breast-feeding 4) Intake of prescription drugs with anti/pro-inflammatory action 5) Intake of prescription drugs with anti/pro-analgesic action 6) Inability to abstain from any anti/pro-inflammatory, or analgesic drugs 48 hours before, or during the study session 7) Inability to obtain at least 6 hours of sleep during the night preceding the study session 8) Known sensitivity or allergy to propranolol or alfentanil 9) Any history of drug or alcohol abuse

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Alfentanil Day 1, Placebo Day 2, and Propranolol Day 3; Alfentanil Day 1, Propranolol Day 2, and Palcebo Day 3: Day 1: Experimental inflammation, and tissue injury sites were created an infusion of alfentanil 100ng/ml was administered over 3 hours.
  Day 2: Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours.
  Day 3: Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump.
  On all study days data were collected to measure inflammation, pain response, and cytokine levels locally.
  Experimental inflammation and tissue injury sites were used for pain testing to determine heat and mechanical pain threshold.
  Interstitial fluid sampling was accomplished with microdialysis. Samples were collected hourly throughout the study day.
  Laser doppler evaluation of tissue perfusion was made at baseline and again at hours 1, 2 and 3 following initiation of the infusions.
- Propranolol Day 1, Placebo Day 2, and Alfentanil Day 3: Day 1: Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours.
  Day 2: Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump.
  Day 3: Experimental inflammation, and tissue injury sites were created an infusion of alfentanil 100ng/ml was administered over 3 hours.
  On all study days data were collected to measure inflammation, pain response, and cytokine levels locally.
  Experimental inflammation and tissue injury sites were used for pain testing to determine heat and mechanical pain threshold.
  Interstitial fluid sampling was accomplished with microdialysis. Samples were collected hourly throughout the study day.
  Laser doppler evaluation of tissue perfusion was made at baseline and again at hours 1, 2 and 3 following initiation of the infusions.
- Placebo Day 1, Propranolol Day 2, and Alfentanil Day 3: Day 1: Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump.
  Day 2: Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours.
  Day 3: Experimental inflammation, and tissue injury sites were created an infusion of alfentanil 100ng/ml was administered over 3 hours.
  On all study days data were collected to measure inflammation, pain response, and cytokine levels locally.
  Experimental inflammation and tissue injury sites were used for pain testing to determine heat and mechanical pain threshold.
  Interstitial fluid sampling was accomplished with microdialysis. Samples were collected hourly throughout the study day.
  Laser doppler evaluation of tissue perfusion was made at baseline and again at hours 1, 2 and 3 following initiation of the infusions.
- Propranolol Day 1, Alfentanil Day 2, and Placebo Day 3: Day 1: Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours.
  Day 2: Experimental inflammation, and tissue injury sites were created an infusion of alfentanil 100ng/ml was administered over 3 hours.
  Day 3: Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump.
  On all study days data were collected to measure inflammation, pain response, and cytokine levels locally.
  Experimental inflammation and tissue injury sites were used for pain testing to determine heat and mechanical pain threshold.
  Interstitial fluid sampling was accomplished with microdialysis. Samples were collected hourly throughout the study day.
  Laser doppler evaluation of tissue perfusion was made at baseline and again at hours 1, 2 and 3 following initiation of the infusions.
- Placebo Day 1, Alfentanil Day 2, and Propranolol Day 3: Day 1: Experimental inflammation and tissue injury sites were created, an infusion of normal saline was administered over 3 hours using a programmable infusion pump.
  Day 2: Experimental inflammation, and tissue injury sites were created an infusion of alfentanil 100ng/ml was administered over 3 hours.
  Day 3: Experimental inflammation and tissue injury sites were created, an infusion of propranolol 30ng/ml was administered over 3 hours.
  On all study days data were collected to measure inflammation, pain response, and cytokine levels locally.
  Experimental inflammation and tissue injury sites were used for pain testing to determine heat and mechanical pain threshold.
  Interstitial fluid sampling was accomplished with microdialysis. Samples were collected hourly throughout the study day.
  Laser doppler evaluation of tissue perfusion was made at baseline and again at hours 1, 2 and 3 following initiation of the infusions.
Period: Overall Study
Arm/Group | Alfentanil Day 1, Placebo Day 2, and Propranolol Day 3 | Propranolol Day 1, Placebo Day 2, and Alfentanil Day 3 | Placebo Day 1, Propranolol Day 2, and Alfentanil Day 3 | Alfentanil Day 1, Propranolol Day 2, and Palcebo Day 3 | Propranolol Day 1, Alfentanil Day 2, and Placebo Day 3 | Placebo Day 1, Alfentanil Day 2, and Propranolol Day 3
Started | 1 | 1 | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alfentanil - Placebo - Propanolol: Participant(s) were randomized to receive an intravenous infusion of alfentanil, normal saline, and propanolol on 3 consecutive study days.
- Propranolol - Placebo - Alfentanil: Participants were randomized to receive an intravenous infusion of propanolol, normal saline, and alfentanil on 3 consecutive study days.
- Placebo - Propanolol - Alfentanil: Participants were randomized to receive an intravenous infusion of normal saline, propanolol, and alfentanil on 3 consecutive study days.
- Alfentanil - Propanolol - Placebo: Participants were randomized to receive an intravenous infusion of alfentanil, propanolol, and normal saline on 3 consecutive study days.
- Propranolol - Alfentanil - Placebo: Participants were randomized to receive an intravenous infusion of propanolol, alfentanil, and normal saline on 3 consecutive study days.
- Placebo -Alfentanil - Propanolol: Participants were randomized to receive an intravenous infusion of normal saline, alfentanil, and propanolol on 3 consecutive study days.
- Total: Total of all reporting groups
Arm/Group | Alfentanil - Placebo - Propanolol | Propranolol - Placebo - Alfentanil | Placebo - Propanolol - Alfentanil | Alfentanil - Propanolol - Placebo | Propranolol - Alfentanil - Placebo | Placebo -Alfentanil - Propanolol | Total
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 2 | 2 | 2 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 0 | 3
  Male | 1 | 1 | 1 | 2 | 0 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Heat Pain Threshold During Infusion in Non-Inflamed Skin
Description: Degrees Centigrade Heat pain was induced with a thermal sensory analyzer (TSA-II, Medoc Advanced Medical Systems, Durham, North Carolina). A thermode was placed in contact with skin on the upper thigh. Starting at a comfortable temperature, the thermode temperature was increased at a measured rate. Study participants pushed a button of a hand-held device at the onset of pain at which point the thermode immediately reduced the temperature. Measurements for analgesia were taken at the sites of non-injured skin. Change form baseline was calculated by subtracting baseline values from the average values obtained 1 and 2 hours after starting the drug infusion.
Time Frame: Participants underwent the pain testing measures at baseline and at 1 and 2 hours after startingthe drug infusion.
Measure: Mean (Standard Deviation); unit: degree centigrade
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
degree centigrade | 1.01 (0.74) | 0.14 (0.26) | 0.01 (0.37)

2. Primary Outcome: Change From Baseline in Heat Pain Threshold During Infusion in Inflamed Skin
Description: Degrees Centigrade Heat pain was induced with a thermal sensory analyzer (TSA-II, Medoc Advanced Medical Systems, Durham, North Carolina). A thermode was placed in contact with skin on the upper thigh. Starting at a comfortable temperature, the thermode temperature was increased at a measured rate. Study participants pushed a button of a hand-held device at the onset of pain at which point the thermode immediately reduced the temperature. Measurements for anti-hyperalgesia were taken at the sites of tissue injury. Change form baseline was calculated by subtracting baseline values from the average values obtained 1 and 2 hours after starting the drug infusion.
Time Frame: Participants underwent the pain testing measures at baseline and at 1 and 2 hours after startingthe drug infusion.
Measure: Mean (Standard Deviation); unit: degrees centigrade
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
degrees centigrade | 3.77 (4.77) | 0.09 (1.31) | -0.28 (0.93)

3. Primary Outcome: Change From Baseline in Mechanical Pain Threshold During Infusion in Non-Inflamed Skin
Description: A metal rod of 0.24 mm diameter mounted onto 10 different weights (1.0, 2.0, 4.1, 8.2,16.3, 20, 32.7,49.0, 65.3, and 81.3g) will be placed perpendicularly onto the skin. Starting with the lightest probe, consecutively heavier probes will be used until a subject reports pain. Subsequently, the same or the next lighter probe will be used if pain is reported for the preceding stimulus, or the same or the next heavier probe will be used if no pain is reported for the preceding stimulus.The procedure will be repeated until seven perceptional changes (painful/non-painful) are registered. Measurements for analgesia were taken at the sites of non-injured skin. Change form baseline was calculated by subtracting baseline values from the average values obtained 1 and 2 hours after starting the drug infusion.
Time Frame: Participants underwent the pain testing measures at baseline and at 1 and 2 hours after startingthe drug infusion.
Measure: Mean (Standard Deviation); unit: weight in grams
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
weight in grams | 10.16 (17.21) | -11.22 (20.65) | -9.53 (18.75)

4. Primary Outcome: Change From Baseline in Mechanical Pain Threshold During Infusion in Inflamed Skin
Description: A metal rod of 0.24 mm diameter mounted onto 10 different weights (1.0, 2.0, 4.1, 8.2,16.3, 20, 32.7,49.0, 65.3, and 81.3g) will be placed perpendicularly onto the skin. Starting with the lightest probe, consecutively heavier probes will be used until a subject reports pain. Subsequently, the same or the next lighter probe will be used if pain is reported for the preceding stimulus, or the same or the next heavier probe will be used if no pain is reported for the preceding stimulus.The procedure will be repeated until seven perceptional changes (painful/non-painful) are registered. Measurements for anti-hyperalgesia were taken at the sites of tissue injury. Change form baseline was calculated by subtracting baseline values from the average values obtained 1 and 2 hours after starting the drug infusion.
Time Frame: Participants underwent the pain testing measures at baseline and at 1 and 2 hours after startingthe drug infusion.
Measure: Mean (Standard Deviation); unit: weight in grams
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
weight in grams | 29.18 (19.86) | -9.07 (7.95) | -11.00 (11.55)

5. Secondary Outcome: TNFα (ng/mL) Change From Baseline During Infusion
Description: TNFα (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 4.92 (6.59) | 5.78 (4.67) | 2.93 (3.36)

6. Secondary Outcome: IL-1β (ng/mL) Change From Baseline During Infusion
Description: IL-1β (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 5.39 (4.89) | 6.99 (6.26) | 7.53 (11.06)

7. Secondary Outcome: IL-2 (ng/mL) Change From Baseline During Infusion
Description: IL-2 (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 2.38 (4.43) | 3.08 (2.52) | 1.65 (1.91)

8. Secondary Outcome: IL-6 (ng/mL) Change From Baseline During Infusion
Description: IL-6 (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 344.2 (414.2) | 214.0 (222.2) | 153.6 (286.6)

9. Secondary Outcome: GMCSF (ng/mL) Change From Baseline During Infusion
Description: GMCSF (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 7.85 (7.77) | 10.75 (5.02) | 6.48 (6.57)

10. Secondary Outcome: IL-8 (ng/mL) Change From Baseline During Infusion
Description: IL-8 (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 486.3 (654.9) | 621.5 (367.0) | 398.7 (422.6)

11. Secondary Outcome: IL-10 (ng/mL) Change From Baseline During Infusion
Description: IL-10 (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 0.35 (1.59) | 0.84 (1.77) | -0.01 (2.03)

12. Secondary Outcome: IL-12 (ng/mL) Change From Baseline During Infusion
Description: IL-12 (ng/mL) was measured in interstitial fluid after collecting samples as follows: Microdialysis catheters (very small, custom-made, sterile, semi-permeable, micro-dialysis catheters) were placed after the 1st laser Doppler measurement. Two catheters were placed at an experimentally inflamed skin site on the left leg. A continuous infusion of sterile 1% albumin solution was started using a programmable pump set at a rate of 2.5µl/min. Samples were collected hourly throughout the remainder of the study day. Samples for analysis were collected before, and 2 and 3 hours after starting the drug infusion. Difference form baseline was calculated by subtracting the baseline concentration form the average concentration determined in samples collected during drug infusion.
Time Frame: Tissue samples were collected at baseline, and 2 and 3 hours after starting the drug infusion.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ng/ml | 2.12 (2.77) | 3.41 (3.58) | 3.38 (4.88)

13. Secondary Outcome: Change in Arbitrary Perfusion Units From Baseline During Drug Infusion
Description: Laser Doppler images were recorded at baseline and at 2 and 3 hours after starting the drug infusion to provide measurements of peripheral blood flow as an objective measure of inflammation. Blood flow was quantified by arbitrary perfusion units. Baseline measurements were subtracted from the average measurements obtained 2 and 3 hours after starting the drug infusion.
Time Frame: Laser doppler images were recorded at baseline and at 2 and 3 hours after starting the drug infusion
Measure: Mean (Standard Deviation); unit: relative flux
Arm/Group | Alfentanil | Propranolol | Placebo
Number analyzed (Participants) | 10 | 10 | 10
relative flux | -234 (191) | -217 (123) | -178 (206)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entire study session on all 3 study days. Collection ended when the participant was discharged.
Description: Adverse events are not reported per intervention as no adverse events were recorded during any intervention.
Groups:
- Alfentanil - Placebo - Propanolol: An infusion of alfentanil 100ng/ml was administered over 3 hours on study 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of normal saline was administered over 3 hours on study 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of propranolol 30ng/ml was administered over 3 hours on study day 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
- Propranolol - Placebo - Alfentanil: An infusion of propranolol 30ng/ml was administered over 3 hours on study day 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of normal saline was administered over 3 hours on study 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of alfentanil 100ng/ml was administered over 3 hours on study 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
- Placebo - Propanolol - Alfentanil: An infusion of normal saline was administered over 3 hours on study 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of propranolol 30ng/ml was administered over 3 hours on study day 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of alfentanil 100ng/ml was administered over 3 hours on study 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
- Alfentanil - Propanolol - Placebo: An infusion of alfentanil 100ng/ml was administered over 3 hours on study 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of propranolol 30ng/ml was administered over 3 hours on study day 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of normal saline was administered over 3 hours on study 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
- Propranolol - Alfentanil - Placebo: An infusion of propranolol 30ng/ml was administered over 3 hours on study day 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of alfentanil 100ng/ml was administered over 3 hours on study 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of normal saline was administered over 3 hours on study 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
- Placebo -Alfentanil - Propanolol: An infusion of normal saline was administered over 3 hours on study 1. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of alfentanil 100ng/ml was administered over 3 hours on study 2. Data were collected to measure inflammation, pain response, and cytokine levels locally.
  An infusion of propranolol 30ng/ml was administered over 3 hours on study day 3. Data were collected to measure inflammation, pain response, and cytokine levels locally.
Arm/Group | Alfentanil - Placebo - Propanolol | Propranolol - Placebo - Alfentanil | Placebo - Propanolol - Alfentanil | Alfentanil - Propanolol - Placebo | Propranolol - Alfentanil - Placebo | Placebo -Alfentanil - Propanolol
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes